CLINICAL TRIAL: NCT00186979
Title: A Phase I Study of ZD1839 (Iressa) in Combination With Irinotecan (Camptosar or CPT-11) and Vincristine in Pediatric Patients With Refractory Solid Tumors
Brief Title: Study of ZD1839 Combined With Irinotecan and Vincristine in Pediatric Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: AstraZeneca (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZD1839
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-10

CONDITIONS: Solid Tumors
Keywords: Refractory Childhood Solid Tumors
MeSH Terms: interventions — Irinotecan; Gefitinib; Vincristine; Cefixime; Cefpodoxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Irinotecan, ZD1839, Vincristine, Cefixime, Cefpodoxime.

INTERVENTIONS:
Drug: Irinotecan, ZD1839, Vincristine, Cefixime, Cefpodoxime. — See Detailed Description section for details of treatment interventions.

SUMMARY:
The purpose of this protocol is to estimate the maximum tolerated dose of gefitinib in combination with fixed dose of irinotecan and vincristine in patients with refractory solid tumors.

DETAILED DESCRIPTION:
Objectives of this study are:

* To determine the dose-limiting toxicities (DLT) of the combination of irinotecan and ZD1839 when given on this schedule.
* To characterize the pharmacokinetics and pharmacodynamics of gefitinib alone and in combination with irinotecan and vincristine.
* To estimate the maximum tolerated dose (MTD) of gefitinib in combination with escalating intravenous irinotecan by using selective intestinal decontamination with oral cefixime or cefpodoxime to prevent diarrhea.
* To estimate the MTD of vincristine (MTD) in combination with gefitinib and irinotecan.

Details of Treatment Interventions

First Cohort:

Standard dose escalation, starting at ZD1839 150 mg/m2/day for 21 days in combination with irinotecan 15mg/m2/day on a daily x 5 for two consecutive week schedule. Dose-limiting diarrhea was seen in this cohort. ZD scheduled was reduced to 12 days. The first dose level (1a) consisted of ZD1839 112.5mg/m2/day for 12 days + irinotecan 15mg/m2/day daily x 5 x 2 and was found to be the MTD in this cohort.

Second Cohort:

Cefixime then added at 4 additional subjects were enrolled at dose level 1c, consisting of ZD1839 at 112mg/m2/day + irinotecan 20mg/m2/day + cefixime 8 mg/kg/day administered once daily, beginning on day -1, and continued to day 14.

Third Cohort:

Irinotecan/ZD1839/Vincristine/Cefixime- Cefixime 8 mg/kg/day administered once daily, beginning on day -1, and continued to day 14, with a maximum dose of 400 mg daily + gefitinib 112.5 mg/m2 orally, daily for 12 days and irinotecan at 15 mg/m2 daily x 5 x 2 +1 mg/m2 (maximum 2mg/dose) on days 1 and 8 with escalating dose of VCR as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 22 years of age.
* Histologic verification of solid tumor malignancy at original diagnosis.
* Has disease considered refractory to conventional therapy or no conventional therapy exists.
* Adequate performance status, bone marrow, liver and kidney function.
* Patients must not have had any previous allergic reactions to penicillin or cephalosporins

Exclusion Criteria:

* Known severe hypersensitivity to ZD1839 or any of the excipients of this product
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's Wort, and CYP3A4 inhibitors
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of trial treatment.
* Incomplete healing from previous oncologic or other major surgery
* Pregnant or breast-feeding
* Patients who have an uncontrolled infection
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded).
* As judged by the investigator, any evidence of uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
* Evidence of any other significant clinical disorder or laboratory finding that makes is undesirable for the subject to participate in the trial.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2003-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | Within the first 30 days of completion of first cycle

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Furman, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Result] A Phase I Study of Gefitinib and irinotecan (IRN) in pediatric patients with refractory solid tumors. WL Furman et al. Vol 22, No 14S (July 15 Supplement), 2004: 8521
- [Result] Effect of Gefitinib on the bioavailability of oral irinotecan in children with refractory solid tumors. K.R. Crews, W.L. Furman, J.C. Panetta, B.B. Freeman, L.C. Iacono, P.J. Houghton, C.F. Stewart. Proceeding of ASCO. Vol 22, No 14S, 2004:2012.
- [Result] Effect of gefitinib on the systemic dispositon of intravenous irinotecan (IRN) in pediatric patients with refractory solid tumors. L.C. Iacono, W.L. Furman, K.R. Crews, J.C. Panetta, B.B. Freeman, N.C. Daw, C.F. Stewart. Proceedings of ASCO. Vol 22, No 14S, 2004:2011.
- See also: St. Jude Children's Research Hospital — http://www.stjude.org